CLINICAL TRIAL: NCT00146198
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Analgesic Efficacy, Safety and Tolerability of ALGRX 4975 in Subjects After Inguinal Hernia Repair
Brief Title: Efficacy and Safety of ALGRX 4975 in Treatment of Postoperative Pain After Hernia Repair
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AlgoRx Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4975-2-007-2; Eudra CT No:2004-004670-88
Record Dates: First submitted 2005-09-04; First posted 2005-09-07 (Estimated); Last update posted 2006-12-20 (Estimated); Status verified 2006-12

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain; Inguinal Hernia Repair; Capsaicin
MeSH Terms: conditions — Pain, Postoperative

INTERVENTIONS:
Drug: ALGRX 4975

SUMMARY:
Hernia repair is one of the most common operations. Whilst there are few complications, pain may last for several weeks and extend the period of convalescence. ALGRX 4975 is an ultra-pure form of capsaicin, which is a pain medicine that has the potential for long-term pain relief following a single administration. This study will determine whether ALGRX 4975 can provide pain relief following hernia repair.

DETAILED DESCRIPTION:
Inguinal hernia correction in adults is one of the most common operations with an annual rate of approximately 2,800 per 1 million people in the United States. Whilst there is little intra and postoperative morbidity, pain may persist for one to several weeks postoperatively and may extend the period of convalescence. ALGRX 4975 is an ultra-pure form of capsaicin, which is a pain medicine that has the potential for long-term pain relief following a single administration. The purpose of this study is to determine whether a single dose of ALGRX 4975, administered by instillation, is able to reduce the postoperative pain following inguinal hernia correction and to evaluate the potential for long term pain relief.

ELIGIBILITY:
Inclusion Criteria:

• The subject has a primary hernia and will undergo hernia repair by standard Lichtenstein mesh repair.

Exclusion Criteria:

* The subject has undergone a lower abdomen surgical procedure in the past.
* The subject is currently scheduled to undergo bilateral inguinal hernia repair.
* Personal or familial contraindications in undergoing general anesthesia.
* Systolic blood pressure greater than 150 mmHg or diastolic greater than 95 mmHg

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-09; Study Completion 2006-02

PRIMARY OUTCOMES:
The average daily VAS pain scores, assessed on a 100 mm VAS during movement upon arising in the morning and retiring in the evening, during the first week after surgery.

SECONDARY OUTCOMES:
Time to supplemental medication usage
Average daily VAS pain scores, assessed during movement upon arising in the morning and retiring in the evening, during the first 4 weeks after surgery
Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Kehlet, MD PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Dagkirurgisk Klinik, Hørsholm, Denmark